CLINICAL TRIAL: NCT02570724
Title: Clinical Effect and Cerebral Vasoconstriction Induced After Epidural Blood Patch Versus Epidural Hydroxyethyl Starch Patch in Patients With Headache Due to Intracranial Hypotension
Brief Title: HES Patch Versus Blood Patch
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5204
Record Dates: First submitted 2015-09-29; First posted 2015-10-07 (Estimated); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Intracranial Hypotension
MeSH Terms: conditions — Intracranial Hypotension | interventions — Hydroxyethyl Starch Derivatives; Blood Patch, Epidural

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Blood Patch arm (Active Comparator): Standard of care arm: injection of autologous blood approximately 40 mL of blood sample into the epidural space at a rate of 1 ml / about 5 seconds.
  Interventions: Biological: blood patch
- Drug: injection of HES " Voluven® " patch arm (Active Comparator): Drug: injection of HES " Voluven® " into the epidural space of 15 to 30 ml at a rate of 1 ml / about 5 seconds
  Interventions: Drug: injection of HES " Voluven® "

INTERVENTIONS:
Drug: injection of HES " Voluven® " — Injection into the epidural space of 15 to 30 ml Voluven ® at a rate of 1 ml / about 5 seconds.
  Other Names: HYDROXYETHYL STARCH
  Arms: Drug: injection of HES " Voluven® " patch arm
Biological: blood patch
  Other Names: injection of autologous blood
  Arms: Blood Patch arm

SUMMARY:
The injection of autologous blood Blood Patch (BP) into the epidural space is the standard treatment for headache associated with intracranial hypotension. It provokes cerebral vasoconstriction. It is cons-indicated in a number of situations (HIV positive, fever, sepsis, leukemia). The purpose of this study is to evaluate another technique using a patch made by injecting an epidural hydroxyethylstarch solution (HES 130, 0.4, 6%) instead of blood patch. This alternative technique is simple to implement and does not have some of the specific blood pressure contra-indications. The study aims at comparing the "Blood Patch" group versus the "HES Patch" in terms of clinical efficacy , tolerance, satisfaction of the anesthetist, ease of implementation and effect of the injection of epidural anesthesia on cerebral blood flow within 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Subjects older than 18 years.·
* Subjects with an intracranial hypertension syndrome secondary to an epidural, spinal or lumbar puncture (and therefore presumed iatrogenic) with a sub arachnoid space or subjects with intracranial hypertension syndrome of primitive origin requiring treatment with epidural Patch ·
* subjects with a temporal window of sufficient quality to carry out the transcranial Doppler ·
* Subjects haven read the informed consent, signed and dated prior to the start of any proceedings related to the tial·
* Subjects affiliated to health insurance·
* Subjects having been informed of the results of a prior medical consultation

Exclusion Criteria:

* Subjects with a cons-indication to an epidural Patch:
* blood disorders constitutional or acquired coagulation with platelets
* Subjects under treatment with curative doses of antiplatelet drugs or anticoagulants
* subjects under shock and / or hypovolemia
* subjects under generalized sepsis or at the puncture site
* any other cons-indication to performing an epidural

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Variation of the pulsatility index (PI) of the middle cerebral artery transcranial Doppler | 36 hours
  Compare the effect of epidural injection of autologous blood (Blood Patch) versus injection of a colloid (HES Voluven ®) on cerebral blood flow.
  this study aims at observing the variation of the pulsatility index (PI) of middle cerebral artery observed by a transcranial Doppler between T0 and 30 minutes after the patch is administered.
  The BP or HEA treatment will be considered equivalent if the proportion of clinical failures and side effects do not differ by more than 5%.

CONTACTS AND LOCATIONS:
Locations (1):
- Service Anesthésie Réanimation Chirurgicale Hôpitaux Universitaires de Strasbourg, 1 avenue Molière, Strasbourg, Strasbourg Cedex, France